CLINICAL TRIAL: NCT01117480
Title: Real Life Evaluation of Rheumatoid Arthritis in Canadians Taking HUMIRA (REACH)
Brief Title: Real Life Evaluation of Rheumatoid Arthritis in Canadians Taking HUMIRA
Acronym: REACH
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: PMOS-CANA-04-01
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Moderate-to-severe Rheumatoid Arthritis
Keywords: Moderate Rheumatoid Arthritis; Rheumatoid Arthritis; Severe Rheumatoid Arthritis; Adalimumab; Clinical Effectiveness
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Moderate-to-severe rheumatoid arthritis: Participants with moderate-to-severe rheumatoid arthritis treated with adalimumab in routine clinical practice

SUMMARY:
The purpose of this study is to evaluate the clinical effectiveness and safety of adalimumab as used in routine clinical practice in adult participants with moderate to severe rheumatoid arthritis (RA) in Canada.

DETAILED DESCRIPTION:
REACH is an observational survey of participants with moderate to severe rheumatoid arthritis taking adalimumab. Participants who volunteer will be asked to provide information about their medical history and experiences with adalimumab. No drug will be provided as a result of participation in the registry. All treatment decisions are independent of participation in the registry.

ELIGIBILITY:
Inclusion Criteria:

* Participant is eligible to take part in the registry as per the product monograph.
* Participants that are naïve to adalimumab therapy / or participants that have been receiving adalimumab therapy for less than 4 months.
* Participant has moderately to severely active RA.
* Participant who has had an inadequate response to one or more Disease Modifying Anti-Rheumatic Drugs (DMARDs).
* Participant received provincial or private (insurance companies) approval for adalimumab.
* Participant is able to give written informed consent and to understand the survey requirements.

Exclusion Criteria:

* Participant to whom a traditional DMARD had never been tried.
* Participant with a known hypersensitivity to adalimumab, or any of its components.
* Participant is receiving free adalimumab as part of a compassionate program or an early access drug distribution program.
* Participant with clinically significant concurrent medical or psychiatric disorders that may influence survey outcomes.
* Participant with any condition that would prevent participation in the survey and completion of the survey procedures including language limitation or possibility that the participant will not be available for a period of time (> 12 months) while being enrolled in the survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate-to-severe rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 1013 (Actual)
Dates: Start 2005-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Assouline, PhD, Study Director — AbbVie Corporation

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate-to-severe Rheumatoid Arthritis
Started | 1013
Completed | 985
Not Completed | 28
Not completed — Protocol Violation | 8
Not completed — Did Not Start Adalimumab Therapy | 20

BASELINE CHARACTERISTICS:
Population: Baseline analyses accounts for Intention to treat (ITT) population (all participants who received at least 1 dose of study drug).
Arm/Group | Moderate-to-severe Rheumatoid Arthritis
Number analyzed (Participants) | 985
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 751
  Male | 234
Disease duration [Mean (Standard Deviation); unit: years] | 10.0 (9.8)
Disease Activity Score 28 (DAS-28) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, erythrocyte sedimentation rate (ESR), and the Subject's Global Assessment of Disease Activity (subject rates disease activity using a likert scale from 0 [low activity] to 10 [high activity]) are included in the DAS28 score. Scores on the DAS28 range from 0 to 10.
  A total of 64 participants had DAS-28 information missing/ unavailable at baseline. These participants were excluded from the efficacy analysis.
  units on a scale | 5.14 (1.60)
Health Assessment Questionnaire (HAQ) [Mean (Standard Deviation); unit: units on a scale] — HAQ-DI is a participant-reported questionnaire referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3); which were summed and averaged to provide an overall score ranging from 0 to 3.
  A total of 13 participants had HAQ information missing/ unavailable at baseline. These participants were excluded from the efficacy analysis.
  units on a scale | 1.39 (0.72)
Rheumatoid Arthritis Disease Activity Index (RADAI) [Mean (Standard Deviation); unit: units on a scale] — The RADAI is a questionnaire used for measuring disease activity. The index consists of 6 questions: (1) global disease activity in the last 6 months, (2) disease activity in terms of current swollen and tender joints, (3) arthritis pain, (4) the current status of health, (5) duration of morning stiffness and (6) tender joints to be rated in a joint list. The RADAI total score is the sum of individual items divided by 5 (range 0-10).
  A total of 13 participants had RADAI information missing/ unavailable at baseline. These participants were excluded from the efficacy analysis.
  units on a scale | 5.4 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Achieved a Disease Activity Score 28 (DAS28) < 2.6
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, erythrocyte sedimentation rate (ESR), and the Subject's Global Assessment of Disease Activity (subject rates disease activity using a likert scale from 0 [low activity] to 10 [high activity]) are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Month 0, 6, 12, 18 and 24
Population: Analyses included all participants who received at least 1 dose of adalimumab (ITT) with baseline data available for DAS-28.
Measure: Number; unit: percentage of participants
Arm/Group | Moderate-to-severe Rheumatoid Arthritis
Number analyzed (Participants) | 921
percentage of participants
  Month 0 | 11
  Month 6 | 13
  Month 12 | 16
  Month 18 | 15
  Month 24 | 16

2. Secondary Outcome: Mean Change From Baseline (Month 0) in Health Assessment Questionnaire (HAQ)
Description: Physical function was evaluated using the Health Assessment Questionnaire - Disability Index (HAQ-DI), a participant-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from baseline in the disability index of the HAQ-DI indicated improvement.
Time Frame: Month 0, 6, 12, 18 and 24
Population: Analyses included all participants who received at least 1 dose of adalimumab (ITT) with baseline data available for HAQ.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Moderate-to-severe Rheumatoid Arthritis
Number analyzed (Participants) | 972
units on a scale
  Month 0 | 1.39 (0.72)
  Month 6 | -0.31 (0.56)
  Month 12 | -0.34 (0.61)
  Month 18 | -0.37 (0.63)
  Month 24 | -0.37 (0.65)

3. Secondary Outcome: Mean Change From Baseline (Month 0) in Rheumatoid Arthritis Disease Activity Index (RADAI)
Description: The RADAI is a questionnaire for participants used for measuring disease activity. The index consists of 6 questions. The items ask the participants about (1) global disease activity in the last 6 months, (2) disease activity in terms of current swollen and tender joints, (3) arthritis pain, (4) the current status of health, (5) duration of morning stiffness and (6) tender joints to be rated in a joint list. The joint list asks about pain in the left and right shoulders, elbows, wrists, fingers, hips, knees, ankles and toes. The first 3 items are all rated on a numeric rating scale from 0 to 10, where higher scores indicate more disease activity. The RADAI total score is the sum of individual items divided by 5 (range 0-10), with a higher score signifying more disease activity.
Time Frame: Month 0, 6, 12, 18 and 24
Population: Analyses included all participants who received at least 1 dose of adalimumab (ITT) with baseline data available for RADAI.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Moderate-to-severe Rheumatoid Arthritis
Number analyzed (Participants) | 972
units on a scale
  Month 0 | 5.4 (2.1)
  Month 6 | -1.55 (2.14)
  Month 12 | -1.77 (2.30)
  Month 18 | -1.88 (2.32)
  Month 24 | -1.93 (2.39)

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the time the participant's informed consent was received until 30 days or 5 half-lives following the intake of the last dose of physician-prescribed treatment i.e., up to 10 weeks.
Description: Non serious adverse events were not collected for this study.
Arm/Group | Moderate-to-severe Rheumatoid Arthritis
Serious Adverse Events (participants affected / at risk) | 43/985
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate-to-severe Rheumatoid Arthritis (N=985)
Leukopenia (Blood and lymphatic system disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Gastric ulcer perforation (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Death (General disorders) | 2
Impaired healing (General disorders) | 1
Appendicitis (Infections and infestations) | 1
Arthritis infective (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Intestinal tuberculosis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 3
Arthritis bacterial (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Angiolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuropathy peripheral (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Cholecystectomy (Surgical and medical procedures) | 1
Coronary artery bypass (Surgical and medical procedures) | 1
Eye operation (Surgical and medical procedures) | 1
Joint arthroplasty (Surgical and medical procedures) | 1
Knee operation (Surgical and medical procedures) | 1
Pharyngeal operation (Surgical and medical procedures) | 1
Spinal fusion surgery (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.